CLINICAL TRIAL: NCT04479293
Title: Assessment of Functional Recovery From COVID-19 Using the Proposed Post- COVID-19 Functional Status Score
Brief Title: Post COVID-19 Functional Status in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU16
Record Dates: First submitted 2020-07-19; First posted 2020-07-21 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COVID-19; Coronavirus Disease; SARS-CoV-2
Keywords: Functional score; Radiologic changes; Psychologic changes; Laboratory; Sleep disturbance
MeSH Terms: conditions — COVID-19; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Post COVID-19 Functional Satus Scale — scale from 0-64 assessing functional limitation

SUMMARY:
Since the outbreak of coronavirus disease - COVID-19 pandemic, most attention has focused on mode of transmission, clinical picture of the disease, treatment and prevention. In the coming weeks and months emphasis will gradually involve the post- acute care of COVID-19 survivors. It is anticipated that COVID-19 may have major impact on physical, cognitive, mental, social health status even in patients with mild disease. Moreover, pulmonary, radiologic, laboratory, sleep issues remain to be addressed

ELIGIBILITY:
Inclusion Criteria:

* All confirmed cases with COVID-19

Exclusion Criteria:

* Non COVID-19 cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed as COVID-19 on clinical, laboratory, radiologic or PCR based are included.
  Patients with different severity mild, moderate, severe , managed at home or in hospitals are included.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
number of functional limitations post COVID-19 | 3-6 month
  scale 0-64 points

SECONDARY OUTCOMES:
number of psychologic changes | 3-6 months
  Hamilton scale, points
Sleep Disturbance and quality | 3-6 months
  ESS scale 0-20, points
Radiologic changes | 3-6 months
  Chest HRCT
Laboratory changes | 3-6 moths
  Complete blood count, C - reactive protein, serum ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Aliae Mohamed-Hussein, MD, Principal Investigator — Assiut University
Locations (1):
- Aliaa Hussein, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided